CLINICAL TRIAL: NCT07308353
Title: Comparative Effects Of Exergaming And Otago Exercise On Anticipatory Postural Control And Sensory Integration In Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/14
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Exergaming; Exercise Therapy; Frail Elderly; Healthy Aging; Mobility Limitation; Muscle Strength; Postural Balance; Proprioception
Keywords: Exergaming; Exercise Therapy; Frail Elderly; Healthy Aging; Mobility limitation; Muscle Strength; Postural Balance; Proprioception
MeSH Terms: conditions — Mobility Limitation | interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otago Exercise Program (Active Comparator): Strengthening exercises
  1. Knee extensor (front knee strength)
  2. Knee flexor (Back knee strength)
  3. Hip abductor (side hip strength)
  4. Ankle plantarflexors (calf raises)
  5. Ankle dorsiflexors (toe raises) Balance retraining exercises
  1. Knee bends 2. Backwards walking 3. Walking and turning around 4. Sideways walking 5. Tandem stance (Heel toe stand) 6. Tandem walk (heel toe walk) 7. One leg stand 8. Heel walking 9. Toe walk 10. Heel toe walking backwards 11. sit to stand 12. Stair walking
  Levels:
  LEVEL A 10 repetitions Hold support LEVEL B 10 repetitions, no support or 10 repetitions, hold support, repeat LEVEL C 10 repetitions No support, repeat LEVEL D 3 x 10 repetitions No support
  Interventions: Procedure: Otago Exercise Program
- Exergaming (Experimental): Games Included:
  20,000 Leaks - multi-directional reaching, internal perturbations Reflex Ridge - anticipatory jumping, ducking, trunk-limb coordination River Rush - dynamic weight shifting, lateral stepping Rally Ball - anticipatory posture control, bilateral upper limb coordination Levels: Basic, Intermediate and Advance
  Interventions: Procedure: Exergaming

INTERVENTIONS:
Procedure: Otago Exercise Program — It will consist of 5 Strengthening Exercises, 12 Progressive Balance Exercises and Walking Training (as tolerated). Protocol will include 3 sessions per week 30 minutes per session for total of 6 weeks Strength exercises will be progressed by increasing repetitions, weight, or duration. Balance tasks will be made challenging by reducing upper limb support, altering base of support, or eyes closing. Progression will be adjusted weekly based on performance and comfort.
  All sessions will be delivered under physiotherapist supervision using the official OEP manual.
  Arms: Otago Exercise Program
Procedure: Exergaming — This intervention involves non-immersive exergaming using the Xbox Kinect system.
  Games Included are 20,000 Leaks, Reflex Ridge, River Rush and Rally Ball. Games will be played 3 times per week for 30 minutes for total of 6 weeks. Three difficulty levels include Basic, Intermediate and Advance. Progression based on participant performance, game scores (gold/silver pins, stars), and therapist observation. For first three weeks 2/3 Game Plays and last three weeks there will be 4/5 game plays.
  Sessions will be supervised one-on-one by a physiotherapist. Participant performance, fatigue, and safety will be monitored throughout the session.
  Arms: Exergaming

SUMMARY:
This study explores whether non-immersive, interactive Exergaming using Xbox Kinect can go beyond conventional exercise by actively training the brain and body to react faster, balance smarter, and move more confidently. Through dynamic games like Reflex Ridge and 20,000 Leaks, we aim to stimulate internal perturbations and real-time Sensory Integration, something Otago doesn't directly target.

In this randomized controlled trial, 36 older adults (aged 55+) will be assigned to either the Exergaming or Otago group. Both groups will receive 6 weeks of supervised balance training (3x/week, 30 mins/session). Primary outcomes include Sensory Integration, measured using modified Clinical Test of Sensory Interaction and Balance (mCTSIB) and Anticipatory postural control assessed through Limits of Stability (LOS) test. Timed up and Go (TUG) will capture functional mobility, which will serve as the secondary outcome in this study.

Both mCTSIB and LOS will be administered using the Postural Stability System of Biodex, a reliable and valid computerized platform designed to objectively quantify postural control under varying sensory conditions.

With evidence-based outcome tools and rigorous analysis, this project doesn't just aim to compare two programs, it's about challenging tradition, modernizing rehab, and making balance training smarter, safer, and more engaging for the elders we serve.

This research could be a leap forward in community-based fall prevention and a step toward a more responsive, personalized future in Neurological Rehabilitation.

DETAILED DESCRIPTION:
Falls are the second leading cause of unintentional injury-related deaths globally and pose as a major public health issue, especially for older individuals. Elderly population experience difficulties in switching quickly between various reliable sensory inputs, which increases risk of falls and injuries. Balance and gait disorders are among the most common causes associated with falls in older individuals. Age-related declines in Sensory Integration and Anticipatory balance responses are one of the leading contributors to falls in older adults.

Rogers et al. in 2021 conducted the only identified head-to-head feasibility RCT directly comparing exergaming interventions with the Otago Exercise Program (OEP) in older adults. This mixed method study establishes the foundational evidence that exergaming and Otago exercise demonstrate comparable clinical benefits on functional balance measures, while identifying need for more detailed comparative studies using objective instrumented measures like Postural Stability System of Biodex.

Chen et al. conducted a comprehensive systematic review and meta-analysis in 2021. This meta-analytic evidence establishes a strong foundation supporting the hypothesis that exergaming interventions can outperform conventional exercise approaches on objective postural control metrics, directly informing the rationale for comparative effectiveness studies examining exergaming versus established fall-prevention programs like the Otago Exercise Program.

The Otago Exercise Program (OEP) is a promising intervention for preventing falls, thereby improving balance and gait. Previous studies reported improved effects on balance using the OEP conducted in a group setting. In 2022 Khumpaneid et al., conducted a study aimed to investigate the effects of a modified-OEP on four components of actual balance (static, dynamic, proactive, and reactive balance) and perceived balance in healthy older adults aged 60-85 years old. The modified-OEP group showed significant improvement in the four components of actual balance and in perceived balance.

The study conducted by Sápi et al., in 2021 aimed to evaluate whether Kinect exergame balance training could beneficially impact sensory reweighting in women over 60 years old. 14 healthy women participated in a single-group pretest/posttest/follow-up usability study. Participants engaged in Kinect for Xbox 360 console games three times a week, for 30 minutes per session, over a 6-week period (18 visits in total). This usability study provides evidence that Kinect exergaming can be a valuable intervention for improving balance and reducing fall risk in older women by enhancing mediolateral stability and sensory reweighting. This implies that the Exergaming may have improved proprioceptive function by providing visual feedback and challenging motor skills.

Pacheco et al., in 2020 conducted a research aimed to evaluate the effectiveness of exergames in improving mobility and balance among older adults without neurological conditions. Exergames led to significant improvements in mobility, as evidenced by better performance on the TUG. The study also found that older adults generally adhered well to exergame programs, with reported adherence rates of up to 100% in some trials.

In this study participants will be randomly allocated in 2 groups, A and B. Each group will contain 18 participants.

Group A will receive Otago Exercise Program Group B will receive treatment through Xbox Exergaming. Otago Exercise Program (OEP) consist of 5 Strengthening Exercises , 12 Progressive Balance Exercises and Walking Training (as tolerated).

Non-immersive exergaming using the Xbox Kinect system, designed to engage multisensory balance responses, anticipatory postural adjustments, and internal perturbation mechanisms through gamified movement. Games Include: 20,000 Leaks, Reflex Ridge , River Rush, Rally Ball.

It is imperative to explore and compare the efficacy of Xbox Kinect-based exergaming versus the Otago Exercise Program in improving sensory integration and anticipatory postural control in older adults. By addressing this research gap, the current study aims to contribute novel insights into the development of more responsive, engaging, and relevant balance interventions for the aging population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 55 years
* Both Genders
* Ambulatory, community-dwelling
* Able to stand unassisted >1 min
* TUG ≤ 13.5 s
* Able to understand and follow command

Exclusion Criteria:

* Diagnosed vestibular and neurological conditions affecting balance
* Orthopedic Conditions i.e., Recent fractures or surgeries, cervical spine issues or severe OA
* Severe visual or auditory deficits
* Use of Assistive device
* Currently enrolled in any other balance or exercise program

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Anticipatory Postural Control | 6 weeks
  It will be assessed using the Limits of Stability test of Postural Stability System (Biodex Balance System). The LOS test measures anticipatory postural control by evaluating the participant's ability to voluntarily shift their center of gravity (COG) toward multiple targets without losing balance. Participants will be instructed to shift their weight toward 8 targets displayed on a screen, using ankle and trunk strategies while standing on a stable platform. Overall LOS Score and Time to complete test will be recorded. Higher values of Overall Directional control indicate better anticipatory balance. Whereas shorter Time to Complete Test reflects quicker anticipatory responses.
Sensory Integration | 6 weeks
  The mCTSIB will be used to assess sensory integration.This test includes the four conditions:
  Eyes Open on Firm Surface, Eyes Closed on Firm Surface, Eyes Open, Foam Surface and Eyes Closed, Foam Surface. Each condition will be tested for 30 seconds, and the system will automatically calculate an overall composite sway score. Higher Sway Index shows lower sensory integration
Functional Mobility | 6 weeks
  The Timed Up and Go (TUG) test will be used to measure functional mobility before and after the intervention. Time to complete (in seconds) will be recorded using a stopwatch. Score ≤13.5 seconds is considered normal for community-dwelling older adults. Score >13.5 seconds indicates reduced functional mobility

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan